CLINICAL TRIAL: NCT07084285
Title: Cervical Facet Injection of Corticosteroids for the Management of Cervicobrachialgia : Protocol for a Randomized Pilot Study
Brief Title: Cervical Facet Injection of Corticosteroids for the Management of Cervicobrachialgia
Acronym: APICALE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APHP220671; 2024-511790-30 (EudraCT Number)
Record Dates: First submitted 2025-07-16; First posted 2025-07-24 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cervicobrachial Neuralgia
Keywords: Neuralgia; cervicobrachialgia; cervicobrachial neuralgia; Foraminal conflict; Posterior intra-articular injection; Cervical spinal injection et corticosteroid
MeSH Terms: conditions — Brachial Plexus Neuritis; Neuralgia | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexamethasone (Experimental): A single dexamethasone injection via the posterior intra-articular route
  Interventions: Drug: Dexamethasone
- Isotonic saline solution (Placebo Comparator): A single isotonic saline solution posterior intra-articular injection
  Interventions: Other: Isotonic saline solution

INTERVENTIONS:
Drug: Dexamethasone — A single 4mg (1mL) dexamethasone injection via the posterior intra-articular route, under CT guidance
  Arms: Dexamethasone
Other: Isotonic saline solution — 1 mL isotonic saline solution, injectable, for a single posterior intra-articular injection, under CT guidance.
  Arms: Isotonic saline solution

SUMMARY:
The main objective is to evaluate the efficacy of a single posterior intra-articular injection of dexamethasone on radicular pain (RP) at 1 month in the treatment of uncomplicated chronic cervicobrachial neuralgia (CBN) in adults, resistant to well-conducted first-line medical treatment.

DETAILED DESCRIPTION:
Cervicobrachial Neuralgia (CBN) is a common condition caused by the compression of a nerve root (C5, C6, C7, or C8) in the cervical spine. In 10% of cases, the duration of symptoms exceeds 3 months, at which point it is considered chronic. Two main etiologies are distinguished :

* Soft disc herniation,
* uncodiscarthrotic foraminal stenosis. The pathophysiology involves both mechanical compression and local inflammation. The initial management is typically medical, provided if there are no signs of severity. If medical treatment fails or if signs of severity are present, surgical intervention is required.

The role of corticosteroid injections in the therapeutic strategy in France remains controversial. Literature on the efficacy of cervical spinal injections is heterogeneous and limited, the safety of such injections is debated, and product availability is restricted.

We hypothesize that posterior intra-articular dexamethasone injection would be effective for radicular pain resistant to first-line medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* Unilateral monoradicular cervicobrachial neuralgia (CBN),
* Predominant radicular pain, with a Radicular Visual Analog Scale (VAS) score ≥ 40/100,
* Imaging (CT or preferably MRI) performed within the last 6 months,
* Foraminal conflict at one level on imaging (CT or preferably MRI) performed within the last 6 months, confirmed by a senior investigator trained in the study,
* Failure of medical treatment that included at least one analgesic (level I to III) and one oral anti-inflammatory (NSAIDs and/or corticosteroids) for at least 7 consecutive days within the last 3 months,
* Discontinuation of oral anti-inflammatory drugs (NSAIDs and/or corticosteroids) 24 hours prior to randomization,
* Current episode duration ≥ 3 months,
* Negative pregnancy test on the day of the procedure for premenopausal female patients,
* Patients of childbearing age must have reliable contraception for the duration of the study,
* Absence of biological inflammatory syndrome, thrombocytopenia, or coagulation disorders on the day of the procedure,
* Patient capable of providing written informed consent prior to participating in the study.

Exclusion Criteria:

* Inability to speak, read, or write French fluently,
* Patient under guardianship or custody, or deprived of liberty,
* No affiliation with social security,
* Neurological signs of severity (clinical motor deficit ≤ 3/5, pyramidal irritation signs, or cervical spinal cord edema on MRI),
* Non-concordant imaging within the last 6 months (absence of conflict, contralateral conflict, or ipsilateral conflict not immediately adjacent), confirmed by a senior investigator trained in the study,
* Recent cervical spine injection (< 3 months),
* Foraminal conflict at more than 2 levels,
* History of cervical spine surgery within the last 12 months or scheduled surgery in this indication within 6 months,
* Secondary CBN (traumatic, infectious, neoplastic, or inflammatory etiology),
* Contraindication to fluoroscopy-guided injection (contrast agent allergy, allergy or contraindication to dexamethasone administration),
* Pregnant women,
* Ongoing participation in another therapeutic trial or interventional research study,
* Patient suspected of non-compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Radicular pain (RP) assessed using a simple self-administered numeric rating scale | Month1
  Simple self-administered numeric rating scale, ranging from 0 (no pain) to 100 (maximum pain), over the 48 hours preceding the 1-month visit assessment.

SECONDARY OUTCOMES:
Cervical pain (numeric rating scale, self-administered) | Day 15, Month1, Month2, Month3
  Numeric rating scale, self-administered, ranging from 0 to 100 over the 48 hours preceding Day 15, 1 month, 2 month and 3 month
Neck Disability Index (NDI) score | Month1 and Month3
  Self-administered functional scale, ranging from 0 to 50 at Month 1 and Month 3
Professional status | Month1 and Month3
  Self-reported : employed, on sick leave, disabled, unemployed, inactive, retired at Month 1 and Month 3
Self-administered EQ5D quality of life scale | Month1 and Month3
Radicular pain (RP) assessed using a simple self-administered numeric rating scale | Over the 48 hours preceding the Day 15, the 2-month and the 3-month visits assessment.
  Simple self-administered numeric rating scale, ranging from 0 (no pain) to 100 (maximum pain), over the 48 hours preceding the visit assessment
The occurrence of adverse events (AEs) and serious adverse events (SAEs) | Day15, Month1, Month2, Month3
The use of analgesics (levels 1, 2, or 3) since the last visit | Day 15, Month1, Month2, Month3
  Self-administered 4-level scale (never, several times a month, several times a week, daily) at Day 15, month1, month2 and 3 months post-injection.

CONTACTS AND LOCATIONS:
Overall Officials: Camille DASTE, MD,PhD, Principal Investigator — AP-HP centre , Université Paris-cité
Locations (1):
- Assistance Publique - Hôpitaux de Paris, Service de Rééducation et de Réadaptation de l'Appareil Locomoteur et des Pathologies du Rachis du Pr François Rannou, Hôpital Cochin, Paris, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No